CLINICAL TRIAL: NCT00515827
Title: A Double-Blind, Randomized, Pilot Study to Measure the Effect of Treatment Intensification With a Potent Integrase Inhibitor, Raltegravir (MK-0518), on the Level of Persistent Plasma Viremia Below 50 Copies/ml in Subjects on Protease Inhibitor- or Non-Nucleoside Reverse Transcriptase Inhibitor-Containing Regimens
Brief Title: Effect of Addition of Raltegravir (MK-0518) to PI- or NNRTI-Based ART Regimens in HIV Infected Subjects With Undetectable Viral Load
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A5244; 10440 (Registry Identifier: DAIDS ES); ACTG A5244
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Raltegravir then Placebo (Arm A) (Experimental): 400 mg raltegravir (MK-0518) administered twice daily in addition to optimized background regimen (OBR) from entry to Week 12; halt raltegravir at Week 12 and add placebo twice daily for 12 weeks
  Interventions: Drug: Raltegravir (MK-0518); Drug: Placebo
- Placebo then Raltegravir (Arm B) (Experimental): Placebo administered twice daily in addition to OBR from entry until Week 12; halt placebo at Week 12 and add 400 mg raltegravir tablet twice daily for 12 weeks
  Interventions: Drug: Raltegravir (MK-0518); Drug: Placebo

INTERVENTIONS:
Drug: Raltegravir (MK-0518) — 400 mg tablet taken orally twice daily
Drug: Placebo — 400 mg placebo tablet taken orally twice daily

SUMMARY:
Raltegravir (MK-0518) is an HIV-1 integrase inhibitor with potent in vitro activity against HIV-1 strains including those resistant to currently available antiretroviral drugs. The purpose of this study is to assess the effectiveness of raltegravir in further reducing viral load in HIV infected patients that have already achieved viral suppression below the level of detection of standard viral load assays when added to antiretroviral therapy (ART).

DETAILED DESCRIPTION:
Although ART has reduced the morbidity and mortality from HIV-1 infection, most individuals who stop ART experience rapid viral rebound. Effective ART can suppress viral load to less than 50 copies/ml; however, current treatment regimens cannot completely eliminate the infection. The primary purpose of this study was to assess the ability of the HIV-1 integrase inhibitor, raltegravir, to reduce viral load when added to ART regimens of HIV-1 infected patients who have achieved viral suppression to less than 50 copies/ml.

The study lasted 24 weeks. Participants were randomly assigned to one of two arms. Participants in Arm A were administered raltegravir in addition to their usual ART regimen from study entry until Week 12. At Week 12, subjects halted raltegravir use and received a placebo until Week 24. Participants in Arm B were administered the placebo in addition to their usual ART regimen from study entry until Week 12. At Week 12, subjects halted the placebo and received raltegravir until Week 24. A real-time polymerase chain reaction (PCR) single copy assay (SCA) capable of detecting 1 copy of HIV RNA was used to assay viral load. The cross-over design allowed assessment of the effect of intensification with raltegravir between the two arms at Weeks 10/12 and every participant enrolled in the study receiving raltegravir for 12 weeks. Primary analysis focused on weeks 10/12 measurement and with no washout period, typical analysis of cross-over design was not intended.

All participants had scheduled visits at Weeks 0, 2, 4, 10, 12, 14, 16, 22, and 24. A targeted physical exam occurred at all visits. Blood and urine collection occurred at selected visits. A medical/medication assessment occurred at trial entry. Drug dispensing and an adherence questionnaire occurred at some visits. A pregnancy test occurred at select visits. Participants' background ART medications were not provided by the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 Infection
* ART for at least 12 months prior to study entry that includes at least two NRTIs and either an NNRTI or a ritonavir-boosted PI
* No change in ART regimen for at least 3 months prior to study entry
* CD4 count of 200 or more at screening
* Viral load below the limit of quantification of an ultrasensitive assay for at least 6 months prior to study entry
* Viral load less than 50 copies/ml using Roche Amplicor HIV-1 RNA Ultrasensitive assay within 60 days of study entry
* All viral load assays obtained within 6 months prior to study entry lower than limits of quantification on all tests
* Pre-ART viral load level greater than 100,000 copies/ml
* Detectable viral load of 1 copy or more on the screening SCA
* Available pre-study entry plasma sample for SCA viral load determination
* Absolute neutrophil count of 750/mm3 or more
* Hemoglobin of 9 g/dL or more for female subjects and 10 g/dL or more for male subjects
* Platelet count of 50,000/mm3 or more
* Calculated creatinine clearance of 30 ml/min or more
* AST, ALT, and alkaline phosphate less than or equal to 5 x ULN
* Total bilirubin less than or equal to 2.5 x ULN. If subject is taking indinavir or atazanavir at screening, total bilirubin must be less than or equal to 5 x ULN.
* Negative serum or urine pregnancy test within 48 hours prior to study entry for females with reproductive potential
* Willing to use acceptable means of contraception

Exclusion Criteria:

* Previous documented virologic failure on an antiretroviral regimen
* Unstable clinical condition that would preclude the subject from undergoing study procedures
* Use of immunosuppressive medications within 60 days prior to study entry. Participants using inhaled or nasal steroids are not excluded.
* Opportunistic infection within 60 days prior to study entry
* Allergy or sensitivity to components of study drug
* Active drug or alcohol abuse
* Serious illness requiring systemic treatment within 60 days prior to study entry
* Receipt of non-HIV vaccination within 30 days prior to study entry
* Receipt of any HIV vaccines
* Plan to change background ART within 24 weeks after study entry
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh T Gandhi, MD, Study Chair — Massachusetts General Hospital; Joseph J Eron Jr., MD, Study Chair — University of North Carolina, Chapel Hill; John W Mellors, MD, Study Chair — University of Pittsburgh Medical Center
Locations (20):
- United States (20):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Cornell CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Harlem ACTG CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - MetroHealth CRS, Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Grinsztejn B, Nguyen BY, Katlama C, Gatell JM, Lazzarin A, Vittecoq D, Gonzalez CJ, Chen J, Harvey CM, Isaacs RD; Protocol 005 Team. Safety and efficacy of the HIV-1 integrase inhibitor raltegravir (MK-0518) in treatment-experienced patients with multidrug-resistant virus: a phase II randomised controlled trial. Lancet. 2007 Apr 14;369(9569):1261-1269. doi: 10.1016/S0140-6736(07)60597-2. PMID 17434401
- [Background] Kassahun K, McIntosh I, Cui D, Hreniuk D, Merschman S, Lasseter K, Azrolan N, Iwamoto M, Wagner JA, Wenning LA. Metabolism and disposition in humans of raltegravir (MK-0518), an anti-AIDS drug targeting the human immunodeficiency virus 1 integrase enzyme. Drug Metab Dispos. 2007 Sep;35(9):1657-63. doi: 10.1124/dmd.107.016196. Epub 2007 Jun 25. PMID 17591678
- [Background] Markowitz M, Morales-Ramirez JO, Nguyen BY, Kovacs CM, Steigbigel RT, Cooper DA, Liporace R, Schwartz R, Isaacs R, Gilde LR, Wenning L, Zhao J, Teppler H. Antiretroviral activity, pharmacokinetics, and tolerability of MK-0518, a novel inhibitor of HIV-1 integrase, dosed as monotherapy for 10 days in treatment-naive HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2006 Dec 15;43(5):509-15. doi: 10.1097/QAI.0b013e31802b4956. PMID 17133211
- [Result] Gandhi RT, Zheng L, Bosch RJ, Chan ES, Margolis DM, Read S, Kallungal B, Palmer S, Medvik K, Lederman MM, Alatrakchi N, Jacobson JM, Wiegand A, Kearney M, Coffin JM, Mellors JW, Eron JJ; AIDS Clinical Trials Group A5244 team. The effect of raltegravir intensification on low-level residual viremia in HIV-infected patients on antiretroviral therapy: a randomized controlled trial. PLoS Med. 2010 Aug 10;7(8):e1000321. doi: 10.1371/journal.pmed.1000321. PMID 20711481
- [Derived] Gandhi RT, Coombs RW, Chan ES, Bosch RJ, Zheng L, Margolis DM, Read S, Kallungal B, Chang M, Goecker EA, Wiegand A, Kearney M, Jacobson JM, D'Aquila R, Lederman MM, Mellors JW, Eron JJ; AIDS Clinical Trials Group (ACTG) A5244 Team. No effect of raltegravir intensification on viral replication markers in the blood of HIV-1-infected patients receiving antiretroviral therapy. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):229-35. doi: 10.1097/QAI.0b013e31823fd1f2. PMID 22083073

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (12 Weeks)
Arm/Group | Raltegravir Then Placebo (Arm A) | Placebo Then Raltegravir (Arm B)
Started | 27 | 26
Completed | 26 | 25
Not Completed | 1 | 1
Not completed — Unwilling to adhere to study requirement | 1 | 1
Period: Second Intervention (12 Weeks)
Arm/Group | Raltegravir Then Placebo (Arm A) | Placebo Then Raltegravir (Arm B)
Started | 26 | 25
Completed | 25 | 25
Not Completed | 1 | 0
Not completed — Consent withdraw | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Then Placebo (Arm A) | Placebo Then Raltegravir (Arm B) | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 24 | 51
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (7) | 49 (11) | 49 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: HIV-1 RNA Level
Description: HIV-1 RNA level, as measured by single copy assay (units are copies/ml), averaged at weeks 10 and 12. The quantification limit of single copy assay was determined by the volume of plasma tested. When averaging the week 10 and 12 measurements, if one of both measurements were below the single copy assay lower limits, the lower limit of quantification was used to compute the average and the result was treated as below the averaged value.
Time Frame: At Weeks 10 and 12
Population: 49 subjects who were on study treatment before week 10 and did not experience virologic failure by week 12
Measure: Median (Inter-Quartile Range); unit: copies/mL
Groups:
- Raltegravir (Arm A): 400 mg raltegravir (MK-0518) administered twice daily in addition to optimized background regimen (OBR) from entry to Week 12
- Placebo (Arm B): Placebo administered twice daily in addition to OBR from entry until Week 12
Arm/Group | Raltegravir (Arm A) | Placebo (Arm B)
Number analyzed (Participants) | 25 | 24
copies/mL | 1.2 [0.4 to 5.0] | 1.7 [0.5 to 2.3]
Statistical Analysis 1: Comparison: Raltegravir (Arm A) vs Placebo (Arm B); Test type: Superiority or Other; p = 0.546, Wilcoxon (Mann-Whitney) — P-value is 2-sided and is not adjusted for multiple comparisons

2. Secondary Outcome: Change in HIV-1 RNA Level
Description: Change in HIV-1 RNA level, as measured by single copy assay (units are copies/ml), from baseline to weeks 10/12 . When averaging the measurements at pre-entry and entry, and at weeks 10 and 12, measurements below the lower limit of quantification (LLQ) were imputed a value of the LLQ divided by 2.
Time Frame: At pre-entry, entry, weeks 10 and 12
Population: All participants who were on study treatment and had not experienced virologic failure
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Raltegravir (Arm A) | Placebo (Arm B)
Number analyzed (Participants) | 25 | 24
copies/mL | -0.2 [-1.2 to 0.2] | -0.1 [-0.6 to 0.4]

3. Secondary Outcome: Change in Total CD4 Cell Count
Description: CD4 cell counts were assessed by flow cytometry at pre-entry and entry (the baseline value was the average of the two measurements) and at week 12
Time Frame: At pre-entry, entry, and week 12
Population: All participants who were on study treatment and had not experienced virologic failure
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Raltegravir (Arm A) | Placebo (Arm B)
Number analyzed (Participants) | 23 | 24
cells/mm^3 | 42 [-52 to 80] | -44 [-117 to 49]

4. Secondary Outcome: Change in Total CD8 Cell Count
Description: CD8 cell counts were assessed by flow cytometry at pre-entry and entry (the baseline value was the average of the two measurements) and at week 12
Time Frame: At pre-entry, entry, and week 12
Population: All participants who were on study treatment and had not experienced virologic failure
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Raltegravir (Arm A) | Placebo (Arm B)
Number analyzed (Participants) | 23 | 24
cells/mm^3 | 55 [-76 to 140] | -39 [-152 to 77]

5. Secondary Outcome: Change in CD4+/CD38+/HLA-DR+ Percent
Description: Level of CD4+ T-cell activation was determined by measuring the percentage of cells that expressed both the activation marker CD38 and Human leukocyte antigen (HLA)-DR. Levels measured at pre-entry and entry were averaged. Change from baseline to week 12 was defined as CD4+/CD38+/HLA-DR+% at week 12 minus CD4+/CD38+/HLA-DR+% at baseline.
Time Frame: At pre-entry, entry, and week 12
Population: All participants who were on study treatment and had not experienced virologic failure
Measure: Median (Inter-Quartile Range); unit: % CD4 cells co-express CD38+ and HLA-DR+
Arm/Group | Raltegravir (Arm A) | Placebo (Arm B)
Number analyzed (Participants) | 20 | 23
% CD4 cells co-express CD38+ and HLA-DR+ | -1 [-2 to 1] | 0 [-1 to 2]

6. Secondary Outcome: Change in CD8+/CD38+/HLA-DR+ Percent
Description: Level of CD8+ T-cell activation was determined by measuring the percentage of cells that expressed both the activation marker CD38 and Human leukocyte antigen (HLA)-DR. Levels measured at pre-entry and entry were averaged. Change from baseline to week 12 was defined as CD8+/CD38+/HLA-DR+% at week 12 minus CD8+/CD38+/HLA-DR+% at baseline.
Time Frame: At pre-entry, entry, and week 12
Population: All participants who stayed on study treatment and had not experienced virologic failures.
Measure: Median (Inter-Quartile Range); unit: % CD8 cells co-express CD38+ and HLA-DR+
Arm/Group | Raltegravir (Arm A) | Placebo (Arm B)
Number analyzed (Participants) | 20 | 23
% CD8 cells co-express CD38+ and HLA-DR+ | -1 [-2 to 2] | 0 [-2 to 5]

7. Secondary Outcome: Number of Participants Who Experienced Study Related Grade 2 or Higher Signs/Symptoms, Grade 3 or Higher Laboratory Abnormalities and Clinical Events From First Day of Treatment to Week 12
Description: Participant who experienced at least one study related grade 2 or higher signs/symptoms, grade 3 or higher laboratory abnormalities and clinical events that are "possibly", "probably" or "definitely" related to study treatment. DAIDS Toxicity Grading Table (2004) was used for grading.
Time Frame: From first day of treatment to week 12
Population: All participants on study treatment
Measure: Number; unit: participants
Arm/Group | Raltegravir (Arm A) | Placebo (Arm B)
Number analyzed (Participants) | 27 | 26
participants | 2 | 0

8. Secondary Outcome: Number of Participants Who Experienced Study Related Grade 2 or Higher Signs/Symptoms, Grade 3 or Higher Laboratory Abnormalities and Clinical Events From Week 12 to Week 24
Description: Participant who experienced at least one study related grade 2 or higher signs/symptoms, grade 3 or higher laboratory abnormalities and clinical events that are 'possibly', probably', or definitely' related to study treatment. DAIDS Toxicity Grading Table (2004) was used for grading.
Time Frame: From week 12 to week 24
Measure: Number; unit: participants
Groups:
- Placebo (Arm A): Placebo administered twice daily in addition to optimized background regimen (OBR) from week 12 to week 24
- Raltegravir (Arm B): 400 mg raltegravir (MK-0518) administered twice daily in addition to OBR from week 12 to week 24
Arm/Group | Placebo (Arm A) | Raltegravir (Arm B)
Number analyzed (Participants) | 23 | 25
participants | 0 | 0

9. Secondary Outcome: Number of Participants Who Discontinued Study Drug
Description: Participants who discontinued randomized study treatment for any reason
Time Frame: From first day of treatment to week 12
Population: All 53 participants
Measure: Number; unit: participants
Arm/Group | Raltegravir (Arm A) | Placebo (Arm B)
Number analyzed (Participants) | 27 | 26
participants | 4 | 1

ADVERSE EVENTS:
Time Frame: From study enrollment until study completion
Description: MedDRA 14
Groups:
- Raltegravir: Baseline to Week 12 for Arm A (Raltegravir then Placebo), and Week 12 to Week 24 for Arm B (Placebo then Raltegravir).
- Placebo: Week 12 to Week 24 for Arm A (Raltegravir then Placebo), and Baseline to Week 12 for Arm B (Placebo then Raltegravir).
Arm/Group | Raltegravir | Placebo
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 10/52 | 16/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Raltegravir (N=52) | Placebo (N=52)
Blood BILirubin increased (Investigations) | 4 | 4
Fatigue (General disorders) | 0 | 3
Pyrexia (General disorders) | 2 | 4
Blood bicarbonate abnormal (Investigations) | 0 | 4
Blood glucose increased (Investigations) | 4 | 5
Dizziness (Nervous system disorders) | 3 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No